CLINICAL TRIAL: NCT01235117
Title: A Phase 2 Study of Azacitidine in Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Azacitidine in Treating Patients With Chronic Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000688119; CTRU-CMML-201; ISRCTN-21428905; EUDRACT-2008-006349-23; LEEDS-HM08/8540; EU-21082
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-11

CONDITIONS: Leukemia
Keywords: chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

INTERVENTIONS:
Drug: azacitidine
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying the side effects of azacitidine and to see how well it works in treating patients with chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and tolerability of azacitidine in patients with chronic myelomonocytic leukemia (CMML).
* To assess the overall response rate in these patients.

Secondary

* To assess the incidence of clinical remission/complete remission or partial response in these patients.
* To assess hematological improvement in patients treated with this drug.
* To assess the overall survival of patients treated with this drug.
* To assess progression-free survival of patients treated with this drug.
* To assess the time to acute myeloid leukemia (AML) transformation of CMML.
* To assess the time to death or AML transformation of CMML.
* To assess the biological correlates.

OUTLINE: This is a multicenter study.

Patients receive azacitidine subcutaneously on days 1-5 and 8-9. Treatment repeats every 4 weeks for at least 6 courses in the absence of loss of response/disease progression or unacceptable toxicity. Patients undergo response evaluation after 6 courses or the last course of treatment. Responders may continue azacitidine until loss of response/disease progression or unacceptable toxicity.

Some patients undergo blood, bone marrow, and buccal swab sample collection periodically for correlative studies.

After completion of study treatment, patients are followed up for 1 month.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * All chronic myelomonocytic leukemia (CMML)-2 patients
  * CMML-1 patients meeting any of the following criteria:

    * Symptomatic bone marrow failure/myeloproliferation defined as any of the following:

      * Red cell transfusion dependence and pre-transfusion hemoglobin < 9.0 g/dL
      * Symptomatic anemia (hemoglobin < 11.5 g/dL)
      * Thrombocytopenia (platelet count < 50 x 10^9/L)
      * Symptomatic bleeding due to platelet functional defect or disseminated intravascular coagulation (DIC)/fibrinolysis
      * White cell count (WCC) > 50 x 10^9/L
    * Düsseldorf Score of intermediate or high risk for proliferative CMML-1 (i.e., WCC > 12 x 10^9/L)
    * International Prognostic Scoring System (IPSS) score of intermediate-2 or high risk for non-proliferative CMML-1 (i.e., WCC < 12 x 10^9/L)
    * Systemic symptoms including weight loss with no alternative explanation (10% of baseline weight within the past 6 months)
    * Symptomatic splenomegaly
    * Symptomatic extramedullary involvement (e.g. skin infiltration or serous effusions)
* No CMML with eosinophilia and 5q33 abnormality

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Creatinine ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative urine pregnancy test
* Fertile patients must use at least 2 forms of effective contraception during study and for 3 months after completion of study therapy
* No other active malignant disease including basal cell or squamous cell carcinoma of the skin
* No known HIV or infectious hepatitis B or hepatitis C
* No active infection
* No known hypersensitivity to azacitidine or mannitol

PRIOR CONCURRENT THERAPY:

* At least 28 days since other prior experimental drug or therapy
* No prior chemotherapy for this disease except hydroxycarbamide
* No other concurrent anticancer or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability
Overall response rate

SECONDARY OUTCOMES:
Incidence of clinical remission/complete remission or partial response according to International Working Group (IWG) criteria
Hematological improvement according to IWG criteria
Overall survival
Progression-free survival
Time to acute myeloid leukemia (AML) transformation of CMML
Time to death or AML transformation of CMML
Biological correlates

CONTACTS AND LOCATIONS:
Overall Officials: David T. Bowen, MD, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (2):
- United Kingdom (2):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland